CLINICAL TRIAL: NCT03052270
Title: "Comparison of Vaginal Progesterone With Arabin Cervical Pessary and Vaginal Progesterone Alone in the Prevention of Preterm Delivery in Singleton Pregnancies With Incidental Premature Shortening of Cervical Length"
Brief Title: Arabin Pessary Combine With Vaginal Progesterone Compare With Vaginal Progesterone Alone to Prevent Preterm Delivery in Singleton Pregnancies
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Former PI Left the Institution
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Mary Stephenson, Professor of Obstetrics and Gynecology, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0599
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Focus: Prevent Preterm Delivery; Incidental Short Cervix at Mid-trimester

STUDY DESIGN:
Intervention Model Description: Randomization between two arms: short cervix with vaginal progesterone and Arabin pessary (study group) versus short cervix with vaginal progesterone alone (control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal progesterone and Pessary (Experimental): 1. Short cervical length equal or less than 20 mm
  2. Singleton pregnant women between 18 -24 weeks with no prior history of preterm deliveries.
  3. 18 years or older at the time of enrollment.
  4. Consent to participate in the study
  Vaginal progesterone as standard of care plus Arabin pessary
  Interventions: Drug: Arabin Pessary
- Vaginal progesterone only (Active Comparator): 1. Short cervical length equal or less than 20 mm
  2. Singleton pregnant women between 18 -24 weeks with no prior history of preterm deliveries.
  3. 18 years or older at the time of enrollment.
  4. Consent to participate in the study
  Vaginal progesterone as standard of care
  Interventions: Drug: Arabin Pessary

INTERVENTIONS:
Drug: Arabin Pessary — Insertion of Arabin pessary for the prevention of preterm delivery

SUMMARY:
1. This will be a randomized prospective and open-label study with no placebo control or blinding of the participants and the research team members. The study is to compare the effectiveness of vaginal progesterone versus combination of vaginal progesterone and Arabin cervical pessary in the prevention of preterm delivery among patients with incidental shortened cervical length.
2. As part of standard clinical care, all pregnant patients usually have cervical length measurements at the mid-trimester during the anatomy scan from 18 to 24 weeks with the GE ultrasound Volusion 8 using the vaginal probe.

   1. Patients with short cervix will be counseled and offered the opportunity to participate in the study.
   2. All participants will be taught how to use the vaginal progesterone once daily prior to bedtime. In addition, those in the combination group will have the cervical pessary placed in the clinic right away or within a week if they request for more time to brood over their diagnosis and weigh on the option of inserting Arabin pessary.
   3. All participants will be followed up in the high-risk obstetric clinic as per standard prenatal care. Frequency of follow up visits will be individualized depending on patient's need and comorbidities. , Participants will be requested to bring the remnant of the vaginal progesterone to the clinic to assess compliance.
   4. Participants in the study will continue their prenatal care with UIC high-risk obstetric clinic until delivery.
   5. The study recruitment will occur for a period of 2 years starting from November 2016 to October 2018 or until all the anticipated numbers of study subjects have been attained.
   6. There will be 10 % over-sampling to cater for those who will drop out from the study or loss to follow up after randomization, and those who delivered in another hospital.
   7. Participants will have access to one of the investigators or the high- risk clinic nurse for any complaints related to their conditions.
   8. Participants can opt out at any stage of the study if they do not want to continue further or if there are any adverse effects.

DETAILED DESCRIPTION:
Preterm birth is the leading cause of neonatal mortality and disability in survivors in the United States. Short cervical length measured by transvaginal ultrasound has been strongly associated with an increased risk of preterm birth. Vaginal progesterone has been proposed as a management option to reduce the risk of preterm birth in asymptomatic women with singleton gestations without prior preterm birth with a very short cervical length. Short cervix in this population is defined as less than or equal to 20 mm, when measured between 18 and 24 weeks.

The American College of Obstetrics and Gynecology (ACOG) and the Society of Maternal Fetal Medicine (SMFM) have proposed the use of vaginal progesterone either micronized progesterone capsule, 200mg daily, or vaginal progesterone gel, 90 mg daily, in asymptomatic women carrying a singleton pregnancy and an incidental finding of short cervix.

Cervical length is usually measured at time of routine anatomical survey fetal between 18 and 24 weeks of gestation for the prevention of preterm birth at less than 37 weeks.

Furthermore, cervical pessary has been used in the prevention of preterm birth for many decades in a few studies with promising results. More recently, the Arabin pessary has been designed with the sole purpose of prevention of preterm birth in pregnant patients with short cervix. It is relatively noninvasive, not operator-dependent and can be easily placed and removed in the outpatient setting.

The purpose of this study is to test the hypothesis that adding the use of the Arabin pessary for women identified with short cervix and undergoing the standard of care treatment with vaginal progesterone, further decreases the risk of preterm birth.

This will be a prospective randomized trial using vaginal progesterone alone compared with the combination of vaginal progesterone and Arabin pessary in the prevention of preterm delivery among women who are incidentally found to have short cervical length. Patients diagnosed with short cervical length with no prior history of preterm deliveries during routine mid-trimester screening will be enrolled in this study and will be randomized into two groups. One group will be given vaginal progesterone only, which is the current standard of care in the United States. The second group will receive Arabin cervical pessary, to be inserted in the clinic at the time of diagnosis, in addition to daily vaginal progesterone.

Vaginal progesterone will be 200 mg or 90 mg of Crinone inserted once daily at bedtime in both groups, depending on patients' insurance coverage. The participants of the study will be followed up in the high risk obstetric clinic as per standard clinic surveillance. They will receive the standard prenatal care and treatment when warranted according to their clinic conditions.

Hypothesis:

The use of Arabin pessary in conjunction with the standard treatment of vaginal progesterone is more effective in reducing preterm deliveries at less than 37 weeks in women identified with short cervix in mid trimester without other risk factors.

Primary Objective:

1. To compare the effectiveness of the combination of vaginal progesterone and Arabin pessary in the prevention of preterm delivery prior to 37 weeks compared to vaginal progesterone alone.

Secondary objectives:

1. Evaluate the rate of preterm delivery prior to 28, 32, 34 weeks in both groups.
2. Evaluate the need for adjunctive interventions such as cervical cerclage, tocolysis, antibiotics and Betamethasone in both groups.
3. To evaluate adverse maternal or fetal outcomes in each study group.
4. Evaluate neonatal intensive care unit admission and composite neonatal morbidity in each study group.

4.0 Eligibility

Participants will be recruited from the investigators' clinical practice if they are diagnosed with short cervical length equal or less than 20 mm at routine ultrasound screening for cervical length during mid-trimester anatomy scan from 18-24 weeks at the UIC ultrasound units. Those with cervical length less than or equal to 20 mm will be randomized (1:1) into two arms: the vaginal progesterone only group and the combined vaginal progesterone and Arabin cervical pessary group. Those with cervical lengths between 20 mm to 25 mm will be followed up in 1 week with repeat transvaginal sonogram, according to the unit protocol but they will be randomized to either group only if they are diagnosed with shorter cervical lengths of 20 mm or less prior to 24 weeks of gestation.

4.1 Inclusion Criteria

1. Short cervical length equal or less than 20 mm
2. Singleton pregnant women between 18 -24 weeks with no prior history of preterm deliveries.
3. 18 years or older at the time of enrollment.
4. Consent to participate in the study

4.2 Exclusion Criteria

1. Previous preterm delivery less than 37 weeks
2. Major fetal anomalies
3. Multiple pregnancy
4. Patient currently with cervical cerclage in-situ for the treatment of incompetence cervix.
5. Regular uterine contractions or significantly dilated cervical canal
6. Age less than 18 years
7. Decline to participate in the study

4.3 Excluded or Vulnerable Populations

Patients who do not have capacity to give consent will be excluded from the study. Women under the age of 18 will not be enrolled in this study.

5.0 Subject Enrollment

1. All pregnant women 18 years old and above who are diagnosed with short cervix during the mid-trimester routine screening for cervical length will be counseled about the treatment options and recruited for the study if they give their consent.
2. They will be recruited at the point of diagnosis of short cervical length at the UIC ultrasound unit or high-risk obstetric clinic in Women Health Center.
3. They will be told that their participation in the study will be voluntary and those already in the study can opt out at any stage if they so desired.
4. Both the participants and those who decline to participate in the study will be treated equally according to their clinical demands. Refusal to participate in the study will not alter in any way the access to other standard of care as the needs arise.
5. All participants will be followed up throughout their pregnancy until delivery. The study enrollment will be from 18 - 24 weeks when they are diagnosed with short cervical length. Final data for each participant will be gathered after delivery.
6. Those with cervical pessary will have the device removed at 37 completed weeks or if they are in labor and any other condition that warrants interruption of the pregnancy. Vaginal progesterone will continue up to 36 completed weeks, as per standard of care.

6.0 Study Design and Procedures

To review, standard prenatal clinical care at UIC includes a cervical length ultrasound evaluation at the time of the routine anatomical fetal survey between 18-24 weeks. When an incidental finding of shortened cervical length is made, patients are typically prescribed vaginal progesterone. They are then followed at the high-risk OB clinic every 2 weeks until delivery. This randomized prospective study compares standard clinical care (vaginal progesterone alone) to standard care plus the Arabin pessary (vaginal progesterone + Arabin cervical pessary) in the prevention of preterm delivery in pregnant women incidentally found to have a significantly shortened cervix between 18 and 24 weeks.

1. This will be a randomized prospective and open-label study with no placebo control or blinding of the participants and the research team members. The study is to compare the effectiveness of vaginal progesterone versus combination of vaginal progesterone and Arabin cervical pessary in the prevention of preterm delivery among patients with incidental shortened cervical length.
2. As part of standard clinical care, all pregnant patients usually have cervical length measurements at the mid-trimester during the anatomy scan from 18 to 24 weeks with the GE ultrasound Volusion 8 using the vaginal probe.

   1. Those with short cervix will be counseled and offered the opportunity to participate in the study.
   2. All participants will be taught how to use the vaginal progesterone once daily prior to bedtime. In addition, those in the combination group will have the cervical pessary placed in the clinic right away or within a week if they request for more time to brood over their diagnosis and weigh on the option of inserting Arabin pessary.
   3. All participants will be followed up in the high-risk obstetric clinic as per standard prenatal care. Frequency of follow up visits will be individualized depending on patient's need and comorbidities. Participants will be requested to bring the remnant of the vaginal progesterone to the clinic to assess compliance.
   4. Participants in the study will continue their prenatal care with UIC high-risk obstetric clinic until delivery.
   5. The study recruitment will occur for a period of 2 years starting from November 2016 to October 2018 or until all the anticipated numbers of study subjects have been attained.
   6. There will be 10 % over-sampling to cater for those who will drop out from the study or loss to follow up after randomization, and those who delivered in another hospital.
   7. Participants will have access to one of the investigators or the high- risk clinic nurse for any complaints related to their conditions.
   8. Participants can opt out at any stage from the study if they do not want to continue further or if there are any adverse effects.

Studies involving use of product

This study uses the Arabin cervical pessary and vaginal progesterone (Endometrin 200 mg or Crinone 90 mg gel).

Arabin cervical pessary:

This is a tissue tolerant non-allergic silicone ring plastic device with a cup-like shape used for cervical insufficiency. It comes in various sizes and it is classified according to its size:

The lower larger diameter (65 or 70 mm) The height (17, 21, 25 or 30 mm) The upper small diameter (32 or 35 mm)

The Arabin cervical pessary can easily be folded and inserted in the upper vaginal around the cervix without pain. The majority of the patients receive a device size of 32 mm of the upper diameter, 21 mm for height and 65 mm for lower diameter. However, participants with significantly funneling of the cervical canal will receive a device of 35 mm of the upper diameter while those with previous vaginal deliveries will receive a device with lower diameter of 70 mm. The length of the vaginal component of the cervix will determine the height of the Arabin pessary to be inserted. Before the applications, participants will be screened and treated for any cervical or vaginal infections. All participants will be screened for bacterial vaginosis, candida infection and Trichomonas, and positive tests will receive appropriate treatments, as per standard of care.

The proposed Arabin cervical pessary will be: Vaginal pessary, CE 0482 MED CERT, EN ISO 13485. Center for Research and Development. Alfred-Herrhausen Str. 44 D 58455 Witten, Germany. Phone: +49 2 302 / 189214. The device will be given to every participant randomized to the pessary group free of charge.

Vaginal pessaries have been used for many years in gynecology for non-surgical treatment of utero-vaginal prolapse and stress urinary incontinence. Different types of pessary based on the indication and the pelvic anatomical defect have been used. Some of the pessaries that have been used in gynecology include: ring, ring with support, Gehrung, Gellhorn, Shaatz, Donut, Cube and inflatable. Vaginal pessaries like Donut and ring with support have been used in pregnancy for the management of cervical insufficiency. However, the pitfall in the use of these pessaries is that they are easily expelled due to the anatomical changes of the vagina in pregnancy that make it difficult for them to fit well in the vagina. With the introduction of Arabin cervical pessary which is designed to allow it wrap around the cervix instead of just placing it in the vagina negate this pitfall. Arabin cervical pessary have been used for many years in Europe for the prevention of preterm delivery in women with cervical incompetence. A Cochrane review by Abdel -Aleem in 2013 showed that Arabin cervical pessary has beneficial effects in reducing preterm birth in women with short cervix, (Abdel-Aleem et al 2013, Liem S et al 2013 and Ting YH et al 2012). This is a non-invasive, and not operator-dependent silicone plastic that is inserted in the vagina to wrap around the cervix thereby preventing it from shortening and dilating. It can easily be placed or removed in an outpatient clinic and it does not require anesthesia. It does not need to be removed for examinations. Premature cervical shortening and dilatation is one of the most important causes of preterm birth. This device does not have systemic adverse effects and the only complaints reported by some of the users is slightly increase vaginal discharge. In another study of systematic review of the efficacy of Arabin cervical pessary, it showed that majority of the patients; > 90 % expressed great satisfaction with the device and they will recommend it to other patients (Sophie M et al 2013).

Endometrin or Crinone vaginal progesterone (Ferring Reproductive Health):

Endometrin (progesterone vaginal insert) is a vaginal insert containing 100 mg of micronized progesterone. Crinone is a vaginal gel (8%) with 90 mg of micronized progesterone. Progesterone is a natural hormone that is often used in pregnancy for various indications. One of the indications is for prevention of preterm deliveries in women with short cervical length. It is usually well tolerated except for some minor side effects such as allergic reactions to some of its components, itching, headache or flushing.

7.0 Expected Risks/Benefits

The expected risks include:

1. If randomized to the pessary group, vaginal erosion of the pessary is possible, but this is extremely rare since the device is soft and with little pressure on the vaginal wall. This has never been an observed side-effect in any patients in investigators clinic that have been using this device for over a year. Moreover, all participants will have access to one of the investigators 24 hours a day and 7 days a week to express any complaints or concerns. In the event that participants feel discomfort with the pessary and they desire to discontinue, the participant will be required to come to the clinic for evaluation and possible removal of the pessary.
2. Allergic reaction to components of vaginal progesterone is also an extremely rare adverse event. The most common sign of allergic reaction is itching. If this occurs, participants will come to the OB ER for immediate evaluation or come to the high risk OB clinic where they will be evaluated and treated accordingly. As vaginal progesterone is prescribed to most women with an incidental finding of shortened cervical length, this risk is no greater than standard clinical care.
3. There is the possibility of increased vaginal discharge from both the daily use of vaginal progesterone and also from the Arabin pessary. While there is also the possibility of infection, this is extremely rare. Participants will be counseled prior to commencement about the possibility of slightly increased vaginal discharge while they are on either or both interventions.
4. There has been report of unsuccessful placement of Arabin pessary. A study done in Belgium in 2013 reported successful placement of Arabin pessary of 82.2 % at first attempt and 90.4 % at second attempt (Cannie MM et al, Ultrasound Obstet Gynecol 2013; 42: 426 - 433). However, the investigators experience with the use of this device at UIC as part of the investigators clinical care has been very encouraging. The investigators have never encountered any unsuccessful attempt at placing the Arabin pessary. This may be largely due to the introduction of a newer version of the device in 2015 which is softer, and more flexible. There are also three different sizes of this device. If any of the investigators encounter difficulty in placing this device in investigator first attempt, it will be withdrawn and the investigator may place the next smaller size of the device. If this is still not successful, the investigator will place the device under direct visualization of the cervix using a vaginal speculum or allow another investigator to attempt placing the device.

ELIGIBILITY:
Inclusion Criteria:

1. Short cervical length equal or less than 20 mm
2. Singleton pregnant women between 18 -24 weeks with no prior history of preterm deliveries.
3. 18 years or older at the time of enrollment.
4. Consent to participate in the study

Exclusion Criteria:

1. Previous preterm delivery less than 37 weeks
2. Major fetal anomalies
3. Multiple pregnancy
4. Patient currently with cervical cerclage in-situ for the treatment of incompetence cervix.
5. Regular uterine contractions or significantly dilated cervical canal
6. Age less than 18 years
7. Decline to participate in the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 57 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Preterm delivery before 37 weeks | 2 years
  1. To compare the effectiveness of the combination of vaginal progesterone and Arabin pessary in the prevention of preterm delivery prior to 37 weeks compared to vaginal progesterone alone.

SECONDARY OUTCOMES:
Preterm delivery before 28 weeks | 2 years
  1. To compare the effectiveness of the combination of vaginal progesterone and Arabin pessary in the prevention of preterm delivery prior to 37 weeks compared to vaginal progesterone alone.
Preterm delivery before 32 weeks | 2 years
  1. To compare the effectiveness of the combination of vaginal progesterone and Arabin pessary in the prevention of preterm delivery prior to 37 weeks compared to vaginal progesterone alone.
Preterm delivery before 34 weeks | 2 years
  1. To compare the effectiveness of the combination of vaginal progesterone and Arabin pessary in the prevention of preterm delivery prior to 37 weeks compared to vaginal progesterone alone.

CONTACTS AND LOCATIONS:
Overall Officials: Mary D Stephenson, MD, MSc, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel-Aleem H, Shaaban OM, Abdel-Aleem MA, Aboelfadle Mohamed A. Cervical pessary for preventing preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2022 Dec 1;12(12):CD014508. doi: 10.1002/14651858.CD014508. PMID 36453699